CLINICAL TRIAL: NCT06665399
Title: Observation Alone for Mild Non-Lactational Mastitis: A Cohort Study.
Brief Title: Observation Alone for Mild Non-Lactational Mastitis
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chen Kai, Vice Director of Dept. of Breast Surgery, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2024-708-01
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Granulomatous Mastitis; Mastitis Chronic
Keywords: Granulomatous Mastitis, Observation, Treatment; Periductal mastitis
MeSH Terms: conditions — Granulomatous Mastitis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observation: In this study, the definition of "observation" is that participants cannot receive the following treatments currently considered to have a clear efficacy for NL-GLM/PDM.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — In this study, the definition of "observation" is that participants cannot receive the following treatments currently considered to have a clear efficacy for NL-GLM/PDM, including surgical treatments (minimally invasive excision or open excision, incision and drainage), ultrasound-guided aspiration, oral corticosteroid therapy, antibiotic treatment, anti-tuberculosis therapy, or ductal lavage therapy. As symptomatic management for pain, the use of NSAIDs is permitted. Additionally, for patients with fistulas or skin lesions, routine wound care is also allowed. These two interventions are not considered as receiving treatment intervention in this study.

SUMMARY:
The goal of this observational study is to investigate the disease progression rate and timing in patients with mild Non-Lactational Granulomatous Lobular / Periductal Mastitis (NL-GLM/PDM) during follow-up with observation alone strategy. The main questions it aims to answer are: What is the rate of disease progression in mild NL-GLM/PDM patients under observation, and what clinical and pathological factors are associated with this progression? Participants with diagnosis of mild NL-GLM/PDM will be monitored over a specified period, with data collected on their clinical outcomes and relevant factors influencing disease progression.

DETAILED DESCRIPTION:
Non-Lactational Granulomatous Lobular / Periductal Mastitis (NL-GLM/PDM) is an inflammatory breast disease of unclear etiology, primarily characterized by the presence of breast masses. A variety of treatment approaches, including intralesional injection, ductal lavage therapy, or corticosteroids had been proposed. Recently, an increasing number of studies have demonstrated that an observation and follow-up strategy for mild cases can yield comparable efficacy. An international consensus recommends that this observation strategy may serve as a first-line treatment approach for mild NL-GLM patients, with additional therapies implemented only upon disease progression.However, in clinical practice, we have observed that some patients with mild NL-GLM/PDM experience disease progression during the observation period, necessitating further treatment. The proportion of this population and the specifics of their disease progression remain unknown. Additionally, the clinical and pathological factors associated with disease progression during observation have not been previously studied. This research aims to conduct a single-center, single-arm, prospective cohort study to investigate the rate and timing of disease progression in mild NL-GLM/PDM during observation, as well as to explore the clinical and pathological factors related to progression. The findings will provide further guidance for subsequent research and clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged 18 to 65 years;
2. Clinically diagnosed with possible non-lactational (more than 6 months since stopping breastfeeding) granulomatous lobular mastitis or periductal mastitis.
3. Mscore ≤ 3 points;
4. Patients with ultrasound findings suggesting localized breast abscess formation must have undergone abscess drainage before enrollment;
5. After education, participants should have a strong willingness for observation and follow-up, and, after discussing with the primary physician, jointly decide to proceed with observation and follow-up;
6. Signed informed consent form.

Exclusion Criteria:

1. Patients with confirmed or suspected breast malignancy;
2. Patients with bilateral mastitis (including those with bilateral simultaneous onset and those with sequential onset of non-lactational granulomatous mastitis);
3. Pregnant patients who are currently in the gestation period;
4. Patients who have had non-lactational mastitis in the same breast within the past year and have undergone treatments such as surgery, oral corticosteroids (for more than 2 weeks), anti-tuberculosis treatment (for more than 2 weeks), or ductal lavage therapy.
5. Patients who received surgery, oral corticosteroids, or anti-tuberculosis treatment for the non-lactational mastitis of the ipsilateral breast within 2 weeks before enrollment.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-lactational mastitis (defined as more than 6 months since stopping breastfeeding) who meet the eligibility criteria at the Breast Tumor Center of Sun Yat-sen Memorial Hospital, Sun Yat-sen University.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
12-weeks Progression Free Proportion | 12 weeks after enrollment
  The proportion of patients who did not experience disease progression events within 12 weeks after enrollment.
12-weeks Treatment Free Proportion | 12 weeks after enrollment
  The proportion of patients who did not experience any predefined treatments within 12 weeks after enrollment.

SECONDARY OUTCOMES:
4-weeks Progression Free Proportion | 4 weeks after enrollment
  The proportion of patients who did not experience disease progression events within 4 weeks after enrollment.
24-weeks Progression Free Proportion | 24 weeks after enrollment
  The proportion of patients who did not experience disease progression events within 24 weeks after enrollment.
4-weeks Treatment Free Proportion | 4 weeks after enrollment
  The proportion of patients who did not experience predefined treatments within 4 weeks after enrollment.
24-weeks Treatment Free Proportion | 24 weeks after enrollment
  The proportion of patients who did not experience predefined treatments within 24 weeks after enrollment.
Median time to progression | 24 weeks after enrollment
  The median time of the first occurrence of a progression event among patients who experience disease progression.
Median time to treatment intervention | 24 weeks after enrollment
  The median time of the first occurrence of a treatment intervention event among patients who experience treatment intervention.

OTHER OUTCOMES:
Correlation between blood test indicators with clinical outcomes | 24 weeks after enrollment
  Explore the correlation between baseline and week 4 inflammatory blood test indicators and their dynamic changes with disease progression and treatment intervention.
Correlation between clinicopathological biomarkers with clinical outcomes | 24 weeks after enrollment
  Explore the correlation between clinical indicators, pathological indicators, and ultrasound indicators at baseline with disease progression and treatment intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Shenshan Medical Center, Sun Yat-sen Memorial Hospital, Shanwei, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided
IPD could be shared if the studies were completed for two years, and approvals were obtained from the administrators.

REFERENCES:
- [Background] Yuan QQ, Xiao SY, Farouk O, Du YT, Sheybani F, Tan QT, Akbulut S, Cetin K, Alikhassi A, Yaghan RJ, Durur-Subasi I, Altintoprak F, Eom TI, Alper F, Hasbahceci M, Martinez-Ramos D, Oztekin PS, Kwong A, Pluguez-Turull CW, Brownson KE, Chandanwale S, Habibi M, Lan LY, Zhou R, Zeng XT, Bai J, Bai JW, Chen QR, Chen X, Zha XM, Dai WJ, Dai ZJ, Feng QY, Gao QJ, Gao RF, Han BS, Hou JX, Hou W, Liao HY, Luo H, Liu ZR, Lu JH, Luo B, Ma XP, Qian J, Qin JY, Wei W, Wei G, Xu LY, Xue HC, Yang HW, Yang WG, Zhang CJ, Zhang F, Zhang GX, Zhang SK, Zhang SQ, Zhang YQ, Zhang YP, Zhang SC, Zhao DW, Zheng XM, Zheng LW, Xu GR, Zhou WB, Wu GS. Management of granulomatous lobular mastitis: an international multidisciplinary consensus (2021 edition). Mil Med Res. 2022 Apr 26;9(1):20. doi: 10.1186/s40779-022-00380-5. PMID 35473758